CLINICAL TRIAL: NCT02473718
Title: Fluid Balance in the ICU - Interventions to Minimize Fluids in Patients With Septic Shock
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201310111
Record Dates: First submitted 2015-06-10; First posted 2015-06-16 (Estimated); Results first posted 2018-03-29 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Septic Shock; Fluid Therapy; Hypotension
MeSH Terms: conditions — Shock, Septic; Hypotension | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fluid minimization group (Experimental): Patients in the fluid minimization arm will have daily fluid intake and output, baseline central venous pressure, mean arterial pressure, central venous oxygen saturation, pulse pressure variation, and inferior vena cava diameters during inspiration and expiration recorded by a dedicated research fellow. Patients who are intubated will also have corrected flow time, stroke volume, cardiac output, and cardiac index recorded via CardioQ. A fluid challenge in the form of a leg raise or infusion of 250 mL of crystalloid over 5 minutes will then be performed and the parameters repeated. The patient will be judged to be fluid responsive or nonresponsive based on the changes in the parameters. Fluid nonresponsive patients will receive the intervention of the fluid minimization protocol by concentrating continuous infusions, discontinuing maintenance fluids, and minimizing carrier fluids. Diuretics and/or ultrafiltration will be utilized to maintain an even to negative fluid balance.
  Interventions: Other: Fluid minimization protocol; Device: Ultrasound
- Usual care group (No Intervention): Patients in the usual care arm will have daily fluid intake and output, baseline central venous pressure, mean arterial pressure, central venous oxygen saturation, pulse pressure variation, and inferior vena cava diameters during inspiration and expiration recorded by a dedicated research fellow. Patients who are intubated will also have corrected flow time, stroke volume, cardiac output, and cardiac index recorded via CardioQ.

INTERVENTIONS:
Other: Fluid minimization protocol — Fluid nonresponsive patients will have continuous infusions concentrated, maintenance fluids discontinued, and carrier fluids minimized. Diuretics and/or ultrafiltration will be utilized to maintain an even to negative fluid balance in patients demonstrating fluid non-responsiveness.
  Arms: Fluid minimization group
Device: Ultrasound
  Arms: Fluid minimization group

SUMMARY:
The purpose of the study is to determine if a protocol that assesses patients' daily fluid intake and output can decrease the overall amount of fluid patients receive during the first five days in the ICU. The study will also determine if decreasing overall fluids can decrease adverse events associated with mechanical ventilation, such as ventilator-associated pneumonias.

The protocol will include daily ultrasounds and blood draws to evaluate fluid balance. Ultrasound will be used to measure changes in the diameter of the inferior vena cava with respiration.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient with septic shock as the primary cause of hypotension
2. Requiring vasopressors for 12 hours after adequate fluid resuscitation and at the time of enrollment

Exclusion Criteria:

1. Patients with a history of end-stage renal disease requiring outpatient dialysis
2. Patients whose goals of care are consistent with comfort measures only
3. Pregnant patients

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

REFERENCES:
- [Background] Alsous F, Khamiees M, DeGirolamo A, Amoateng-Adjepong Y, Manthous CA. Negative fluid balance predicts survival in patients with septic shock: a retrospective pilot study. Chest. 2000 Jun;117(6):1749-54. doi: 10.1378/chest.117.6.1749. PMID 10858412
- [Background] Angus DC, Linde-Zwirble WT, Lidicker J, Clermont G, Carcillo J, Pinsky MR. Epidemiology of severe sepsis in the United States: analysis of incidence, outcome, and associated costs of care. Crit Care Med. 2001 Jul;29(7):1303-10. doi: 10.1097/00003246-200107000-00002. PMID 11445675
- [Background] Dellinger RP, Levy MM, Rhodes A, Annane D, Gerlach H, Opal SM, Sevransky JE, Sprung CL, Douglas IS, Jaeschke R, Osborn TM, Nunnally ME, Townsend SR, Reinhart K, Kleinpell RM, Angus DC, Deutschman CS, Machado FR, Rubenfeld GD, Webb SA, Beale RJ, Vincent JL, Moreno R; Surviving Sepsis Campaign Guidelines Committee including the Pediatric Subgroup. Surviving sepsis campaign: international guidelines for management of severe sepsis and septic shock: 2012. Crit Care Med. 2013 Feb;41(2):580-637. doi: 10.1097/CCM.0b013e31827e83af. PMID 23353941
- [Background] Michard F, Boussat S, Chemla D, Anguel N, Mercat A, Lecarpentier Y, Richard C, Pinsky MR, Teboul JL. Relation between respiratory changes in arterial pulse pressure and fluid responsiveness in septic patients with acute circulatory failure. Am J Respir Crit Care Med. 2000 Jul;162(1):134-8. doi: 10.1164/ajrccm.162.1.9903035. PMID 10903232
- [Background] Michard F, Teboul JL. Predicting fluid responsiveness in ICU patients: a critical analysis of the evidence. Chest. 2002 Jun;121(6):2000-8. doi: 10.1378/chest.121.6.2000. PMID 12065368
- [Background] Marik PE, Baram M, Vahid B. Does central venous pressure predict fluid responsiveness? A systematic review of the literature and the tale of seven mares. Chest. 2008 Jul;134(1):172-8. doi: 10.1378/chest.07-2331. PMID 18628220
- [Background] Marik PE, Baram M. Noninvasive hemodynamic monitoring in the intensive care unit. Crit Care Clin. 2007 Jul;23(3):383-400. doi: 10.1016/j.ccc.2007.05.002. PMID 17900477
- [Background] Rivers E, Nguyen B, Havstad S, Ressler J, Muzzin A, Knoblich B, Peterson E, Tomlanovich M; Early Goal-Directed Therapy Collaborative Group. Early goal-directed therapy in the treatment of severe sepsis and septic shock. N Engl J Med. 2001 Nov 8;345(19):1368-77. doi: 10.1056/NEJMoa010307. PMID 11794169
- [Background] Vincent JL, Sakr Y, Sprung CL, Ranieri VM, Reinhart K, Gerlach H, Moreno R, Carlet J, Le Gall JR, Payen D; Sepsis Occurrence in Acutely Ill Patients Investigators. Sepsis in European intensive care units: results of the SOAP study. Crit Care Med. 2006 Feb;34(2):344-53. doi: 10.1097/01.ccm.0000194725.48928.3a. PMID 16424713
- [Background] National Heart, Lung, and Blood Institute Acute Respiratory Distress Syndrome (ARDS) Clinical Trials Network; Wiedemann HP, Wheeler AP, Bernard GR, Thompson BT, Hayden D, deBoisblanc B, Connors AF Jr, Hite RD, Harabin AL. Comparison of two fluid-management strategies in acute lung injury. N Engl J Med. 2006 Jun 15;354(24):2564-75. doi: 10.1056/NEJMoa062200. Epub 2006 May 21. PMID 16714767
- [Derived] Chen C, Kollef MH. Targeted Fluid Minimization Following Initial Resuscitation in Septic Shock: A Pilot Study. Chest. 2015 Dec;148(6):1462-1469. doi: 10.1378/chest.15-1525. PMID 26291900

RESULTS

PARTICIPANT FLOW:
Groups:
- Fluid Minimization Group: Patients in the fluid minimization arm will have daily fluid intake and output, baseline central venous pressure, mean arterial pressure, central venous oxygen saturation, pulse pressure variation, and inferior vena cava diameters during inspiration and expiration recorded by a dedicated research fellow. Intubated patients will also have corrected flow time, stroke volume, cardiac output, and cardiac index recorded via CardioQ. Fluid challenge as a leg raise or infusion of 250 mL of crystalloid over 5 minutes will be performed and parameters repeated. Fluid responsiveness based on the changes in the parameters. Fluid nonresponsive patients will undergo the fluid minimization protocol.
  Fluid minimization protocol: Fluid nonresponsive patients will have continuous infusions concentrated, maintenance fluids discontinued, and carrier fluids minimized. Diuretics and/or ultrafiltration will be utilized to maintain an even to negative fluid balance.
Period: Overall Study
Arm/Group | Fluid Minimization Group | Usual Care Group
Started | 41 | 41
Completed | 41 | 41
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluid Minimization Group | Usual Care Group | Total
Number analyzed (Participants) | 41 | 41 | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 31 | 62
  >=65 years | 10 | 10 | 20
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 58 [45 to 65] | 60 [50 to 68] | 58 [51 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 20 | 41
  Male | 20 | 21 | 41
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 41 | 41 | 82
APACHE II score [Median (Inter-Quartile Range); unit: units on a scale] — Acute Physiology And Chronic Health Evaluation II (APACHE II) score is a severity of illness scoring system. An integer score from 0 to 71 is calculated based on physiologic parameters within the first 24 hours of admission to the ICU. Higher scores correspond to more severe disease and an increasing risk of death.
  units on a scale | 25 [22 to 28.5] | 26 [20.5 to 30] | 25 [21.5 to 29.5]
SOFA score [Median (Inter-Quartile Range); unit: units on a scale] — Sequential organ failure assessment (SOFA) score is a severity of illness scoring system. An integer score from 0 to 24 is calculated based on physiologic parameters at the time of admission. Higher scores correspond to more severe disease and an increasing risk of death.
  units on a scale | 13 [11 to 15] | 12 [11 to 15] | 13 [11 to 15]
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 32.62 [24.37 to 37.85] | 31.13 [25.98 to 37.41] | 32.33 [24.84 to 37.85]
Intubation status [Count of Participants; unit: Participants] | 28 | 31 | 59
Presence of ARDS [Count of Participants; unit: Participants] | 26 | 25 | 51
Presence of COPD [Count of Participants; unit: Participants] | 5 | 7 | 12
Presence of hypertension [Count of Participants; unit: Participants] | 14 | 19 | 33
Presence of hyperlipidemia [Count of Participants; unit: Participants] | 10 | 10 | 20
Presence of diabetes mellitus [Count of Participants; unit: Participants] | 12 | 10 | 22
Presence of systolic heart failure [Count of Participants; unit: Participants] | 4 | 5 | 9
Presence of diastolic heart failure [Count of Participants; unit: Participants] | 4 | 4 | 8
Presence of chronic kidney disease [Count of Participants; unit: Participants] | 6 | 3 | 9
Presence of active malignancy [Count of Participants; unit: Participants] | 16 | 10 | 26
Presence of end-stage liver disease [Count of Participants; unit: Participants] | 13 | 7 | 20

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Fluid Administered
Description: Cumulative volume of crystalloid boluses, continuous infusions, and colloid fluids administered in mL by day 3
Time Frame: Day 3
Population: Five patients in the fluid minimization group and two patients in the usual care group died prior to the first time point analysis at day three. One patient in the usual care group was transferred out of the ICU prior to the first time point analysis at day 3.
Measure: Median (Inter-Quartile Range); unit: mL of study fluid
Arm/Group | Fluid Minimization Group | Usual Care Group
Number analyzed (Participants) | 36 | 38
mL of study fluid | 4417 [3139 to 6528] | 4110 [2702 to 10004]

2. Primary Outcome: Cumulative Fluid Administered
Description: Cumulative volume of crystalloid boluses, continuous infusions, and colloid fluids administered in mL by day 5
Time Frame: Day 5
Population: Five patients in the fluid minimization group and four patients in the usual care group died prior to analysis at day 5. Five patients in the fluid minimization group and six patients in the usual care group were transferred out of the ICU prior to analysis at day 5.
Measure: Median (Inter-Quartile Range); unit: mL of study fluid
Arm/Group | Fluid Minimization Group | Usual Care Group
Number analyzed (Participants) | 31 | 31
mL of study fluid | 6244 [5106 to 8497] | 8690 [4211 to 13197]

3. Primary Outcome: Net Fluid Balance
Description: Difference between cumulative volume of all IV fluids administered and all outputs in mL by day 3
Time Frame: Day 3
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Fluid Minimization Group | Usual Care Group
Number analyzed (Participants) | 36 | 38
mL | 1952 [48 to 5003] | 3124 [767 to 10103]

4. Primary Outcome: Net Fluid Balance
Description: Difference between cumulative volume of all IV fluids administered and all outputs in mL by day 5
Time Frame: Day 5
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Fluid Minimization Group | Usual Care Group
Number analyzed (Participants) | 31 | 31
mL | 2641 [-1837 to 5075] | 3616 [-1513 to 9746]

5. Secondary Outcome: Ventilator Days
Description: Number of days requiring mechanical ventilation support, including continuous noninvasive positive pressure ventilation
Time Frame: Hospital stay, median of 16 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Fluid Minimization Group | Usual Care Group
Number analyzed (Participants) | 41 | 41
days | 8 [3.25 to 15.25] | 5 [3 to 9]

6. Secondary Outcome: Rate of Renal Replacement Therapy
Description: Percentage of patients requiring renal replacement therapy
Time Frame: ICU stay, median of 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Fluid Minimization Group | Usual Care Group
Number analyzed (Participants) | 41 | 41
Participants | 17 | 16

7. Secondary Outcome: Mortality
Description: Percentage of patients who died during their hospitalization
Time Frame: Hospital stay, median of 16 days
Measure: Count of Participants; unit: Participants
Arm/Group | Fluid Minimization Group | Usual Care Group
Number analyzed (Participants) | 41 | 41
Participants | 23 | 20

8. Secondary Outcome: Mortality
Description: Percentage of patients who died during their ICU stay
Time Frame: ICU stay, median of 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Fluid Minimization Group | Usual Care Group
Number analyzed (Participants) | 41 | 41
Participants | 23 | 20

ADVERSE EVENTS:
Time Frame: Hospital length of stay, median of 16 days
Arm/Group | Fluid Minimization Group | Usual Care Group
All-Cause Mortality (participants affected / at risk) | 23/41 | 20/41
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/41
Other Adverse Events (participants affected / at risk) | 0/41 | 0/41

LIMITATIONS AND CAVEATS:
Pilot study with small sample size Single center study Possible undetected crossover effect or Hawthorne effect

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No